CLINICAL TRIAL: NCT03945864
Title: The Use of Antimicrobial Synthetic Bone Grafts in the Treatment of Bone Infection
Brief Title: Antimicrobial Synthetic Bone Grafts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, NUSRET KOSE, Professor of Orthopedics and Traumatology, Eskisehir Osmangazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-2491
Record Dates: First submitted 2019-03-31; First posted 2019-05-10 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Bone Infection; Bone Graft Infection

STUDY DESIGN:
Intervention Model Description: experimental group will be compared with parental antibiotics group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antimicrobial synthetic bone graft (Experimental): This group will have parenteral antibiotics and antimicrobial (silver ions) synthetic bone graft
  Interventions: Device: antimicrobial synthetic bone graft
- parenteral antibiotics with pure synthetic bone graft (Active Comparator): This group will have parenteral antibiotics and pure synthetic bone graft
  Interventions: Device: parentaral antimicrobials and pure bone grafts

INTERVENTIONS:
Device: antimicrobial synthetic bone graft — It will be determined whether the silver ion-doped antimicrobial synthetic bone graft that has the capacity to fill the bone voids also has the capacity to treat the infection in the bone in 12 patients with chronic osteomyelitis
  Arms: antimicrobial synthetic bone graft
Device: parentaral antimicrobials and pure bone grafts — Historical data of the department will be used for comparison of the results
  Arms: parenteral antibiotics with pure synthetic bone graft

SUMMARY:
This project aims to produce synthetic bone tissue graft that supports bone regeneration and combats infection simultaneously, according to industry standards and regulations. This original and high value added biomaterial "silver doped calcium phosphate based synthetic bone tissue " will be used in clinical trials in patients with osteomyelitis and implant-related infections for the treatment.

Chronic bone infections are one of the most important problems in orthopedic surgery and are not just a problem of developed societies. When open fracture cases, which may get infected in 1-50%, implant-related infections and diabetic foot ulcer cases are taken into consideration, osteomyelitis will be seen as a very common problem all over the world. Multiple surgeries, long-term use of antibiotics and the high costs affects all societies. The use of synthetic bone grafts is growing faster than the natural bone grafts in the world. USA has spent 246 million US dollars for the use of synthetic bone graft in 2010. For the treatment of bone infections antibiotic impregnated synthetic bone grafts with different characteristics are used. Although these antibiotic impregnated synthetic bone grafts are superior compared to antibiotic bone cement with the implementation of different antibiotics and to be absorbable but they cannot show optimum benefit because the release of antibiotics is not due to host matrix degradation but diffusion control. The other issue to be considered as this regard that the development of microbial resistance to these antibiotics which is also a serious problem. Innovative synthetic bone graft with better contribution of the needs of mechanical properties, depending on the applied bone region, optimized antimicrobial activity and bone tissue regeneration are needed.

In this study, it will be determined whether this silver ion -doped antimicrobial synthetic bone graft that has the capacity to fill the bone voids that may occur in chronic bone infection during disease process or after surgical debridement, also has the capacity to treat the infection in the bone will be used in 12 patients who had been diagnosed as chronic osteomyelitis to see if it cause any unwanted side effect in normal usage conditions and generates unacceptable risks. Clinical, laboratory and radiological investigations will be used to demonstrate the healing of the infections and the cavities in the bone. Blood and urine levels of silver will be detected from patients.

Antimicrobial activity of silver is well-known. The effectiveness of the silver and potential toxicity is related to the dose of silver and application form. In orthopedics, the use of silver is mostly limited to elemental silver coating of metal implants. There is no biotechnologic approach manufactured silver ion -doped calcium phosphate -based synthetic bone graft in the health sector yet. Ionic silver has advantages such as low toxicity, no tolerance of silver against bacteria, and strong antibacterial activity. The trapping of silver ions in the calcium phosphate based ceramic structure overcomes the other systems with its controlled release and its ability to be effective at minimum doses. The project is an original work since it will contribute to bone regeneration while at the same time removing the infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic osteomyelitis, infected non-union or implant-associated infection with an indication for artificial bone grafting who read and accept the Informed consent.
* Male and female patients older than 18 years
* Patients without heart, lung, renal or hepatic failure, epilepsy, cerebrovascular attack or ischemia
* Patients who are not allergic to antibiotics
* Patients with additional immunosuppression such as malignancy, diabetes mellitus, poly travma and open fractures
* Patients using oral or parenteral corticosteroids, methotrexate, cyclosporine or other immunosuppressive drugs

Exclusion Criteria:

* Patients who have not accepted the method.
* Patients outside the working age range
* Pregnant women
* Patients with heart, lung, renal, hepatic failure, epilepsy, cerebrovascular attack or ischemia
* Patients with allergy to antibiotics
* Patients with another silvery implant in the body like a silver-coated implant
* Patients with a history of known allergies or hypersensitivity to silver

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
bony healing of the cavities in the bone | 12 months
  Number of Participants with bony healing of the cavities in the bone by x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the publication of the study nidividual participant data (IPD) will be available to other researchers.